CLINICAL TRIAL: NCT03244774
Title: Phase I Study of the Combination of Apatinib and POF (Paclitaxel Plus Oxaliplatin Plus 5-fluorouracil Plus Leucovorin)
Brief Title: Phase I Study of the Combination of Apatinib and POF
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNF 007
Record Dates: First submitted 2017-07-29; First posted 2017-08-10 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — apatinib; Paclitaxel; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apatinib plus POF (Experimental): This study will include a sequential evaluation of 3 subjects per cohort. Cohort 1: apatinib 250 mg per day and POF. Cohort 2: apatinib 375 mg per day and POF. Cohort 3: apatinib 500 mg per day and POF. Cohort 4: apatinib 625 mg per day and POF. Cohort 5: apatinib 750 mg per day and POF.
  A dose limiting toxicity (DLT) event is defined as any of the following events in the first 4-week period:
  1. CTCAE Grade 4 event (except for neutropenia lasting for ≤ 5 days);
  2. Grade 3 non-hematologic toxicity (except for nausea and vomiting that could be improved with optimal supportive care, escalation of alkaline phosphatase)
  If a DLT is experienced in any cohort, the cohort will be expanded to 6 subjects. If 2 DLTs are experienced in any cohort, the dose escalation ceased. The MTD was defined as the dose having at most two out of six patients experience DLT.
  Interventions: Drug: Apatinib; Drug: POF

INTERVENTIONS:
Drug: Apatinib — Apatinib 250mg p.o. qd in first cohort (3 subjects). 375mg p.o. qd in second cohort (3 subjects). 500mg p.o. qd in third cohort (3 subjects). 625mg p.o. qd in forth cohort (3 subjects); 750mg p.o. qd in fifth cohort (3 subjects).
  Other Name:
  Other Names: YN968D1
Drug: POF — The POF regimen consisted of a 3-hour infusion of paclitaxel (135 mg/m2) followed by oxaliplatin (85 mg/m2) and Calcium Levofolinate (200 mg/m2).Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days.
  Other Names: Paclitaxel plus Oxaliplatin plus Luecovorin plus 5-Fluorouracil

SUMMARY:
In previous studies, we found that POF (A combination of oxaliplatin, fluorouracil and Paclitaxel) regimen appears to be of good efficacy and is well tolerated in patients with advanced gastric cancer. Apatinib is an orally antiangiogenic agent. It was approved and launched in China in 2014 as a 3rd-line treatment for patients with advanced gastric cancer. Therefore, investigators initialize this dose escalation phase I study to explore the safety of combination of apatinib and POF as first-line treatment for advanced gastric cancer. Investigators will analyze the maximum tolerated dose (MDT) and dose-limiting toxicity (DLT) of apatinib in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced unresectable, histologically confirmed adenocarcinoma of the gastric or gastroesophageal junction.
2. No previous treatment with chemotherapy or radiation therapy.
3. Ability to take medications orally.
4. With or without measurable lesions.
5. Patients must have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.
6. Without serious system dysfunction and could tolerate chemotherapy. With normal marrow, liver and renal function: a hemoglobin (HGB) of ≥100g/L (without blood transfusion during 14 days); a leucopenia count of ≥4.0×109/L; a platelet count of ≥100×109/L; a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL); a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault); a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL or ≤5 UNL in case of liver metastasis.
7. Life expectancy ≥3 months.
8. With normal electrocardiogram results and no history of congestive heart failure.
9. Without bleeding and thrombosis disease.
10. With normal coagulation function: activated partial thromboplastin time (APTT), prothrombin time (PT) and INR, each ≤ 1.5 x ULN.
11. Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug
12. With written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.
13. With good compliance and agree to accept follow-up of disease progression and adverse events.

Exclusion Criteria:

1. Patients with a history of another neoplastic disease within the past three years, excluding basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer.
2. Patients with brain or central nervous system metastases, including leptomeningeal disease.
3. Pregnant (positive pregnancy test) or breast feeding.
4. Serious, non-healing wound, ulcer, or bone fracture.
5. Significant cardiac disease as defined as: unstable angina, New York Heart Association (NYHA) grade II or greater, congestive heart failure, history of myocardial infarction within 6 months Evidence of bleeding diathesis or coagulopathy.
6. History of a stroke or CVA within 6 months.
7. Clinically significant peripheral vascular disease.
8. Inability to comply with study and/or follow-up procedures.
9. Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | From enrollment to completion of study. Estimated about 12 months.
  Dose limiting toxicity (DLT) is referred to grade 3 non-hematological toxicity or grade 4 hematological toxicity according to NCI CTCAE 4.03 criteria
Maximum tolerance dose | From enrollment to completion of study. Estimated about 12 months.
  Maximum tolerance dose (MTD) is the dose of treatment in the cohort where there are 2 cases of DTL reported.

SECONDARY OUTCOMES:
Objective response rate | From enrollment to 3 months after treatment
  Clinical response of treatment according to RESIST v1.1 criteria (ORR, objective response rate).
Progression-free survival | From enrollment to progression of disease. Estimated about 6 months.
  The length of time from enrollment until the time of progression of disease (PFS, progression-free survival).
Overall survival | From enrollment to death of patients. Estimated about 1 year.
  The length of time from enrollment until the time of death (OS, overall survival).

CONTACTS AND LOCATIONS:
Overall Officials: Rongbo Lin, Principal Investigator — Fujian Cancer Hospital
Locations (1):
- Rongbo Lin, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No